CLINICAL TRIAL: NCT03865303
Title: Acute Care Learning Laboratory-Reducing Threats to Diagnostic Fidelity in Critical Illness
Brief Title: Learning Lab for Diagnostic Fidelity
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian W. Pickering, M.B., B.Ch., Pricinple Investigator, Mayo Clinic
Other Study IDs: 18-007115; R18HS026609 (AHRQ)
Record Dates: First submitted 2019-01-04; First posted 2019-03-06 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Critical Illness
Keywords: Critical Illness; Patient Safety; Delivery of Health Care; Electronic Health Records
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diagnostic error and delay remain a leading cause of preventable harm and death in the United States. Using a learning laboratory structure, researchers will implement mixed-methods research approaches to identify the systemic weaknesses that contribute to diagnostic error and delay in the hospital setting. The knowledge gained from research innovative will allow researchers to design, develop, implement, and refined a suite of human-centered tools that can be deployed to reduce the risk of diagnostic error and delay in both community and academic hospital settings.

DETAILED DESCRIPTION:
Despite the recognition that diagnostic errors an delays are a major contributor to preventable deaths in the USA, little progress has been made to reduce mortality outcomes from this known killer. An effective strategy leading to meaningful reduction in diagnostic error and delay rates has not made its way into practice. This proposal is unique and novel and combines mixed-methods research approaches with systems engineering research approaches to understand the interplay of the multiple factors contributing to diagnostic error and delay. The knowledge gained from this holistic approach will then be used within the learning laboratory to inform the design, development, evaluation, and refinement of the solutions to diagnostic error and delay. "Control Tower" will be the staging ground for the in situ learning laboratory and will be built on top of a well-established clinical informatics infrastructure and hospital environment open to innovation and practice change.

ELIGIBILITY:
Inclusion Criteria

* For EMR review all adults admitted to the hospital ages 18 and older with research authorization
* For survey-clinicians including physicians, advanced care practitioners
* For focus groups and interviews-clinicians including physicians, advanced care practitioners

Exclusion Criteria

* Age <18 years old
* No research authorization
* Refusal to give consent

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. All patients at risk of diagnostic error will be eligible for the study.
  2. We will include both sexes and all genders and all minority populations as they present with the risk of diagnostic error in the hospitals.
  Given the nature of the study, which focuses on patients with or at risk of diagnostic error, outreach efforts to underrepresented populations or individuals would not be possible.
Sampling Method: Non-Probability Sample
Enrollment: 25551 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Validation of automated phenotypes | 1 year
  Use data from the patient electronic medical record to identify the number of diagnostic error or delay to validate clinical environment automated phenotypes
Adoption (Number of time the Control Tower used during the clinical encounters) | 1 year
  Standardized process tracking sheets to track each time the control tower system is triggered and used.
Implementation Acceptability | 1 year
  Focused questions about beliefs, attitudes, usability by healthcare providers

CONTACTS AND LOCATIONS:
Overall Officials: Brian W Pickering, M.B., B.Ch., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Health System - Mankato MCHS, Mankato, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials